CLINICAL TRIAL: NCT02468687
Title: A Phase I, Open Label Dose Escalation Trial of Orally Administered N-methyl-pyrrolidone (NMP) in Patients With Relapsed or Refractory Myeloma
Brief Title: NMP in Relapsed / Refractory Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREC/14/MH/159
Record Dates: First submitted 2015-06-02; First posted 2015-06-11 (Estimated); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Multiple Myeloma
Keywords: Relapsed/Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — N-methylpyrrolidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- N-methyl-pyrrolidone (Other): NMP dose escalation in accelerated phase and standard phase
  Interventions: Drug: N-methyl-pyrrolidone

INTERVENTIONS:
Drug: N-methyl-pyrrolidone — NMP will be taken each morning as a single daily dose of oral suspension at a concentration of 50mg/ml on an empty stomach at least 30 minutes prior to food.
  Other Names: NMP

SUMMARY:
The study will evaluate if the N-methyl-pyrrolidone (NMP) can be safely administered to humans at doses, which induce measurable immunological and anti-tumour effects in patients with myeloma who are resistant to or intolerant of lenalidomide and bortezomib.

DETAILED DESCRIPTION:
N-Methyl-2-pyrrolidone (NMP) is a small molecule acetyl-lysine mimetic compound with potent (low micromolar range) immunomodulatory and direct anti-myeloma activity attributable to BETbromodomain inhibition at higher concentrations. NMP is nontoxic, stable and already in use as a solvent in biomedical applications. It has been the subject of numerous toxicity studies in humans and been demonstrated to have few adverse effects. The study is proposing an empiric starting dose of 50mg daily, 50% of that seen in healthy volunteers with no observable toxicity. Dose escalation will follow a rule based on accelerated trial design in order to minimise the number of patients treated at sub-therapeutic doses and minimise the length of the study. During the accelerated dose-escalation phase, one patient will be entered per cohort with a dose escalation increment of 100%, with up to 6 dose escalation and up to two dose de-escalation levels.The accelerated phase ends when one patient experiences DLT during the first cycle of treatment or when a total of two patients have experienced moderate toxicity during the first cycle of treatment regardless of the dose level; or the most recent patient has been treated at the highest dose level in the first cycle. If 1 patient experiences a DLT in the first cycle at any dose level, the cohort will be further expanded to a total of 6 patients treated at the same dose level. The maximum tolerated dose (MTD) in the study will be defined as the highest dose in which the incidence of DLT was less than 33%.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of plasma cell myeloma defined by WHO 2008 criteria
2. Measurable disease as defined by at least one of:

   * serum M protein ≥5g/L
   * urine M protein ≥ 200mg/24hrs
   * involved serum free light chain ≥ 100mg/L
   * measurable (by imaging at the discretion of the investigator) soft tissue plasmacytoma
3. Relapsed, refractory or intolerant of both bortezomib and lenalidomide

Definitions:

* refractory at least 4 weeks of therapy administered, with less than a partial response by IMWG criteria
* relapsed from previous response (PR or greater) to therapy, with subsequent disease progression as defined as development of bone marrow dysfunction (fall in Hb of 20g/L or platelet count <100 x 109/L) due to increased bone marrow plasmacytosis
* OR new lytic bone lesions
* OR increase in serum M protein of 5g/L
* OR absolute increase of involved serum free light chain of >250mg/L
* intolerant: grade 2 or higher toxicity unresponsive to dose adjustment 4. Prior autologous stem cell transplant, unless ineligible for transplant by the discretion of the investigator.

  5. age ≥18 years 6. ECOG performance status <2 7. The following values within 7 days of commencing NMP (blood transfusions prior to study entry are permitted)
* Haemoglobin >80g/L
* Absolute neutrophil count >1.0 x 109/L
* Platelet count ≥ 25 x 109/L
* Creatinine clearance >30ml/min (by Cockcroft/Gault)
* Bilirubin ≤ 3x upper limit of normal (ULN)
* ALT ≤ 3 x ULN
* Left ventricular ejection fraction (LVEF) ≥45% (by gated cardiac blood pool scan or echocardiography) 9. Life expectancy > 3 months 10. Able to give written informed consent 11. In the opinion of the investigator, willing and able to comply with required study procedures 12. Able to take oral medications (no malabsorptive condition)

Exclusion Criteria:

1. Pregnant or breastfeeding female patients
2. Female of child bearing potential unwilling or unable to use two methods of contraception
3. Received chemotherapy, immunotherapy or biological therapy within two weeks of enrolment. Prednisolone up to 20mg per day permitted for non-myeloma indications.
4. Patients with a history of another malignancy within 2 years of the baseline visit, excluding treated non-melanotic skin cancer and in-situ carcinoma.
5. Patients with known CNS involvement unless previously treated and well controlled for a period of ≥3 months AND which do not require the use of steroids.
6. Uncontrolled intercurrent illness including, but not limited to:

   * Active or uncontrolled infection, including active HIV or viral (A, B or C) hepatitis. NOTE: Patients with controlled infection on antibiotic or antifungal therapy are eligible i.e. the patient should be afebrile for at least 72 hours and be haemodynamically stable.
   * Impaired cardiac function, including any of the following:

     * Myocardial infarction within previous 3 months prior to starting study
     * Symptomatic congestive heart failure (New York Heart Association Class III, IV)
     * Symptomatic coronary artery disease
     * Cardiac arrhythmia not controlled by medication
     * Clinically significant resting bradycardia (<50 beats per minute)
     * Long QT syndrome or a known family history of long QT syndrome or QTc > 450 msec on baseline ECG (using the QTcF formula). If QTcF >450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc
     * Inability to monitor the QT/QTc interval on ECG
     * Other clinically significant uncontrolled heart disease (e.g. unstable angina or uncontrolled hypertension)
   * Impaired hepatic or renal impairment (see inclusion criteria)
   * Uncontrolled diarrhoea, nausea or vomiting
7. concomitant exposure to another investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Adverse events to establish the Maximum Tolerated Dose (MTD) | 28 days
  Each patient will be monitored for adverse events during the first cycle of NMP treatment (28 days) to establish the maximum tolerated dose

SECONDARY OUTCOMES:
Optimum biological dose (OBD) | 6 months
  The maximum changes in correlative biomarkers will be tested at the specific time-points. Descriptive statistics will be used to analyse data from correlative studies and summarized in graphical or tabular formats as appropriate.
Safety of the repeated dosing of NMP by oral administration - possible toxicities | 6 months
  To assess safety, the numbers and rates (with confidence intervals) of patients experiencing any haematological and non-haematological and specific grade 3+ adverse events experienced at each given dose level and schedule of NMP will be calculated, over the full treatment period and by cycle
Pharmacokinetic properties of NMP after oral administration | Predose,0.5,1,2,4,8, 24 hours post dose
  Pick plasma concentrations (Cmax) of NMP
Response rate measured using IMWG criteria | 6 months up to 2 years
  Patients will be evaluated for response after every 28 day cycle for the first 6 cycles of treatment and thereafter every 2 months in follow up using the IMWG criteria for multiple myeloma.
Time to progression from start of treatment | up to 3.5 years
  Patients will be assessed for disease progression weekly in Cycle 1, then monthly on D1 of each cycle during treatment for the first 6 months and then monthly until disease progression, next anti-cancer treatment or death. Time to progression from start of treatment will be estimated using Kaplan Meier survival curves.

CONTACTS AND LOCATIONS:
Overall Officials: David Ritchie, Prof, Principal Investigator — Melbourne Health
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia